CLINICAL TRIAL: NCT06845020
Title: The Effects of CSF of Patients with Glioblastomas on the Microglial Immune Profile
Brief Title: CSF Proteomic Characterization of Glioblastomas
Status: Not yet recruiting | Type: Observational
Sponsor: Univeridad Autonoma de Guadalajara (Other)
Collaborators: Mayo Clinic (Other); Hospital Valentin Gomez Farias (Other)
Responsible Party: Principal Investigator, Maria G. Zavala-Cerna, Director of Research Development in Health Sciences, Univeridad Autonoma de Guadalajara
Other Study IDs: T05-273-1324-4794-19-00
Record Dates: First submitted 2025-01-31; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-01

CONDITIONS: Glioblastoma; Glioblastoma WHO Grade IV; Glioblastoma (GBM); Glioblastoma Multiforme of the Brain; Glioblastoma, Adult
Keywords: Glioblastoma; Cerebrospinal fluid; CSF; GBM; Proteomics; Biomarker
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid, tumor tissue and blood serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with definitive diagnosis of glioblastoma: The cohort includes patients with a histopathological diagnosis of glioblastoma, defined by the 2021 guidelines: IDH-Wildtype diffuse and astrocytic glioma in adults
  + microvascular proliferation or necrosis OR + TERT promotor mutation OR + EFGR gene amplification OR + +7/-10 chromosome copy number changes.

SUMMARY:
The goal of this observational study is to identify proteins that can be found in the cerebrospinal fluid (CSF) of patients with grade IV brain tumors, specifically glioblastomas, and correlate these proteins with progression free survival, overall survival and performance status (functionality). All participants with high probability of glioblastoma will initially be included, final inclusion will be dependent on the definitive histopathological diagnosis of the tumor.

The main question is:

Can the researchers identify a proteomic profile in CSF from study participants with glioblastoma in association with a longer progression free survival? Participants will undergo the following procedures, that do not deviate from normal standard diagnostic care.

1. Lumbar puncture to obtain CSF.
2. Blood draw.
3. Trans-surgical tissue sample of the brain tumor. Additionally participants will be planned for follow up appointments every 3 months following the first 12 months after the surgical tumor resection.

DETAILED DESCRIPTION:
To successfully complete the study the following procedures will be implemented after obtaining informed consent:

1. Serum blood sample acquisition and storage
2. CSF sample acquisition Of all subjects included in the study a CSF sample will be taken. The sampling will be pre-surgical by lumbar puncture. Before the lumbar puncture all patients will undergo brain imaging (CT or MRI), as well as an fundoscopic exam and a blood draw. Through patient history and clinical examination other neurological pathology is discarded (neurological focalization, altered mental status, recent seizures or any other previous or recent neurological pathology). Patients with lumbar puncture contraindications as sampling method will undergo trans-surgical sampling, as initial procedure performed during surgery to avoid contamination. All sampling must be taken before any radio- and/or chemotherapy.
3. Storage of sampled CSF The CSF sample obtained will be minimally 3 mL (3 tubes of 1 mL), in sterile tubes without any type of additives. The sample will be stored at -80 °C.
4. Tumour tissue acquisition and storage Of all subjects included in the study, tumour tissue samples will be obtained from the central zone, posteriorly molecular analysis and identification of coding genes for significant proteins in CSF will be performed with MALDI-TOF.

After obtaining the patient background information and the tissue samples (CSF, tumour and serum) genetic and histological testing will be performed to obtain glioblastoma diagnosis, following current guidelines, the next parameters must be present for definitive glioblastoma diagnosis, and thus inclusion in the study:

1. IDH-Wildtype diffuse and astrocytic glioma in adults

+ microvascular proliferation or necrosis OR + TERT promotor mutation OR + EFGR gene amplification OR + +7/-10 chromosome copy number changes. When definitive diagnosis is obtained and inclusion in this study is confirmed there will be programmed follow-up visits at 3, 6, 9 and 12 months, where a previously designed questionnaire similar to the admission questionnaire will be performed to specify patient evolution, and functionality current adjuvant treatment, additionally a full physical exam including neurological exam will be performed, with a radiological imaging study (CT or MRI). In case of decease, this will be closely registered by contacting the patient or family one week before the follow-up appointment to confirm the appointment, in case of deceasement date and cause must be registered.

Statistical Analysis:

For the descriptive phase of the statistical analysis, it is intended to use the mean and standard deviation for the variables with parametric distribution and the median with Interquartile range for the variables with non-parametric distribution. Qualitative variables such as protein identification will be reported in frequencies and percentages. The inferential phase includes the creation of contingency tables and chi square. For the analysis of progression-free survival and overall survival, Kaplan Meier curves will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of glioblastoma (histopathological and molecular).
* Patients who voluntarily accept participation in this study.
* Patients aged 18 or older.

Exclusion Criteria:

* Patients who cannot be followed up at the Regional Hospital 'Dr. Valentin Gomez Farias' ISSSTE.
* Contamination of the required sample (CSF, serum, tumor).
* Patients with whom no sampling was obtained or subjects with incomplete background information.
* Patients who decide to withdraw participation from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population includes patients who arrive at the Hospital Regional 'Dr. Valentin Gomez Farias' ISSSTE, who have a high probability of glioblastoma diagnosis, based on clinical presentation and imaging. Additionally the population includes 5 patients whose samples and information has already been stored at the Mayo Clinic Florida.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Measured at 3, 6, 9, and 12 months, after participant recruitment.
  The length of time the participants are still alive after tumor resection (initial recruitment date), including disease progression.

SECONDARY OUTCOMES:
Progression free survival | Measured at 3, 6, 9, and 12 months, after participant recruitment.
  Progression free survival is defined by the amount of time the patient lives with glioblastoma from the start of treatment (surgical resection) without progression of disease.
  Progression of disease is defined as follows: an increase in tumor size, or; new cancerous lesiones on imaging, or; a non-measurable increase of malignant disease (eg.: paraneoplastic syndrome).
Performance status | Measured at baseline, 3, 6, 9, and 12 months, after participant recruitment.
  The Karnofsky performance status (KPS) will be used to measure the functionality of patients with cancer, and their ability to perform daily tasks. This be used this as a measurement of disease progression and to correlate different KPS with the proteomics found. The KPS scale measures patients performance on a scale from 0 to 100% with 10% intervals, 0% meaning patient deceased and 100% normal activity, without signs of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Guadalupe Zavala Cerna, MD, PhD, Principal Investigator — Universidad Autónoma de Guadalajara; Hugo Guerrero Cazares, MD, PhD, Study Chair — Mayo Clinic Jacksonville, Florida.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmid D, Warnken U, Latzer P, Hoffmann DC, Roth J, Kutschmann S, Jaschonek H, Rubmann P, Foltyn M, Vollmuth P, Winkler F, Seliger C, Felix M, Sahm F, Haas J, Reuss D, Bendszus M, Wildemann B, von Deimling A, Wick W, Kessler T. Diagnostic biomarkers from proteomic characterization of cerebrospinal fluid in patients with brain malignancies. J Neurochem. 2021 Jul;158(2):522-538. doi: 10.1111/jnc.15350. Epub 2021 Apr 9. PMID 33735443
- [Background] Skog J, Wurdinger T, van Rijn S, Meijer DH, Gainche L, Sena-Esteves M, Curry WT Jr, Carter BS, Krichevsky AM, Breakefield XO. Glioblastoma microvesicles transport RNA and proteins that promote tumour growth and provide diagnostic biomarkers. Nat Cell Biol. 2008 Dec;10(12):1470-6. doi: 10.1038/ncb1800. Epub 2008 Nov 16. PMID 19011622
- [Background] Schuhmann MU, Zucht HD, Nassimi R, Heine G, Schneekloth CG, Stuerenburg HJ, Selle H. Peptide screening of cerebrospinal fluid in patients with glioblastoma multiforme. Eur J Surg Oncol. 2010 Feb;36(2):201-7. doi: 10.1016/j.ejso.2009.07.010. Epub 2009 Aug 11. PMID 19674866
- [Background] Jayaram S, Gupta MK, Polisetty RV, Cho WC, Sirdeshmukh R. Towards developing biomarkers for glioblastoma multiforme: a proteomics view. Expert Rev Proteomics. 2014 Oct;11(5):621-39. doi: 10.1586/14789450.2014.939634. Epub 2014 Aug 13. PMID 25115191
- [Background] Kohata T, Ito S, Masuda T, Furuta T, Nakada M, Ohtsuki S. Laminin Subunit Alpha-4 and Osteopontin Are Glioblastoma-Selective Secreted Proteins That Are Increased in the Cerebrospinal Fluid of Glioblastoma Patients. J Proteome Res. 2020 Aug 7;19(8):3542-3553. doi: 10.1021/acs.jproteome.0c00415. Epub 2020 Jul 16. PMID 32628487
- [Background] Hori T, Sasayama T, Tanaka K, Koma YI, Nishihara M, Tanaka H, Nakamizo S, Nagashima H, Maeyama M, Fujita Y, Yokozaki H, Hirose T, Kohmura E. Tumor-associated macrophage related interleukin-6 in cerebrospinal fluid as a prognostic marker for glioblastoma. J Clin Neurosci. 2019 Oct;68:281-289. doi: 10.1016/j.jocn.2019.07.020. Epub 2019 Jul 18. PMID 31327593
- [Background] Miller AM, Shah RH, Pentsova EI, Pourmaleki M, Briggs S, Distefano N, Zheng Y, Skakodub A, Mehta SA, Campos C, Hsieh WY, Selcuklu SD, Ling L, Meng F, Jing X, Samoila A, Bale TA, Tsui DWY, Grommes C, Viale A, Souweidane MM, Tabar V, Brennan CW, Reiner AS, Rosenblum M, Panageas KS, DeAngelis LM, Young RJ, Berger MF, Mellinghoff IK. Tracking tumour evolution in glioma through liquid biopsies of cerebrospinal fluid. Nature. 2019 Jan;565(7741):654-658. doi: 10.1038/s41586-019-0882-3. Epub 2019 Jan 23. PMID 30675060
- [Background] Carrano A, Zarco N, Phillipps J, Lara-Velazquez M, Suarez-Meade P, Norton ES, Chaichana KL, Quinones-Hinojosa A, Asmann YW, Guerrero-Cazares H. Human Cerebrospinal Fluid Modulates Pathways Promoting Glioblastoma Malignancy. Front Oncol. 2021 Mar 4;11:624145. doi: 10.3389/fonc.2021.624145. eCollection 2021. PMID 33747938